CLINICAL TRIAL: NCT03838952
Title: The Efficacy of Traditional Chinese Herbal Medicine for Dementia: a Pilot Study
Brief Title: The Efficacy of Traditional Chinese Herbal Medicine for Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-07-021B
Record Dates: First submitted 2019-02-01; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Chinese Herbal Medicine; Herbal treatment
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Phytotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese herbal medicine group (Experimental): drug for the subjects
  Interventions: Drug: Herbal medicine

INTERVENTIONS:
Drug: Herbal medicine — Each pack: Jia Wei Xiao Yao San granule(5 gm), Gou Teng granule (1.1 gm),and Ba Ji Tian (1.1 gm), 2 times per day for 12 weeks.

SUMMARY:
The Clinical trial is a pilot study for treatment of Alzheimer dementia by traditional Chinese herbal medicine(TCM).

DETAILED DESCRIPTION:
Dementia is a chronic, progressive neurodegenerative syndrome, characterized by an abroad category of non-reversible impairment in cerebral function, making a long-term and gradually decrease in the ability to mental cognitive tasks and performance of daily activities.

The World Health Organization says that 47.5 million people around the world are living with dementia. Alzheimer's disease is the most common type of dementia. Alzheimer's disease is often getting worse with time, affecting memory, language, and thought.

According to the record from Ministry of Health and welfare in Taiwan. The population over 65 year-old is more than 3.36 million. It is estimated that there are more than 250,000 people with mental disabilities, and nearly 600,000 people with mild cognitive impairment (MCI). Alzheimer's disease is accounting for 60-70%, the most common type of dementia. With the aging of population, experts predict that the number of patients suffering from Alzheimer's disease will be up to 800,000.

In 2016, a study based on the health insurance database in Taiwan showed that 78.2% of patients will take Chinese medical treatment, such as herbal medicine, acupuncture or traumatology medical therapy like massage after diagnosed as Alzheimer's disease during 1997-2008.

The clinical trial is a pilot study. The main purpose of this study is to evaluate the efficacy of traditional Chinese herbal medicine(TCM) of Alzheimer's dementia. The participants diagnosed as Alzheimer's dementia will be given Traditional Chinese herbal medicine powder, each pack included of Jia Wei Xiao Yao San granule(5 gm), Gou Teng granule (1.1 gm),and Ba Ji Tian (1.1 gm), 2 times per day for 12 weeks. The participants will be assessed by the MMSE, IADL, NPI-Q, GDS, QOL-AD, CCMQ, which will be conducted at baseline, 0weeks, 12weeks, and follow-up (16 weeks). To see if the traditional Chinese herbal medicine can improve the symptoms of Alzheimer's dementia or its related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of mild to moderate Alzheimer dementia;
2. aged over 65 years old in both gender;
3. MMSE score between 14 and 26;
4. adequate vision and hearing ability to complete all study tests;
5. with a stable caregiver.

Exclusion Criteria:

1. a medical history of other dementia types, like Frontotemporal dementia, Dementia with Lewy Bodies, Vascular Dementia, and mixed type, et al;
2. known of other neurological diseases, cranial nervous system cancer
3. severe liver or kidney dysfunction (alanine aminotransferase>200 IU/L, aspartate transaminase>200 IU/L or serum creatinine >2.5 mg/dl);
4. severe cardiovascular disease (heart failure, coronary heart disease)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-11 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Mini-Mental State Examination(MMSE) | week 0, 12, 16
  Global cognition will be assessed by the MMSE,which will be conducted at baseline, 0weeks, 12weeks, and follow-up (16 weeks).
Changes of Instrumental Activities of Daily Living (IADL) | week 0, 12, 16
  The instrumental activities of daily living (IADL) contains 8 items ,such as shopping, cooking, doing laundry, handling finances, using telephone, mode of transportation, responsibility for own medication and housekeeping.The IADL wil be conducted baseline, 12weeks, and follow-up (16 weeks)
Changes of Neuropsychiatric Inventory(NPI-Q) | week 0, 12, 16
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is an informant-based instrument that measures the presence and severity of 12 Neuropsychiatric Symptoms (NPS) in patients with dementia, as well as informant distress. The NPI-Q will be conducted at baseline, 12 weeks, and follow-up (16 weeks).
Changes of Geriatric Depression Scale (GDS) | week 0, 12, 16
  The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly, which will be conducted at baseline, 12weeks, and follow-up (16 weeks).

SECONDARY OUTCOMES:
Blood test (AST/ALT/Serum Creatinine) | week 0, 16
  Check liver and kidney function through blood test at baseline, and follow-up (16 weeks).
Changes of Quality of Life-Alzheimer's Disease (QOL-AD) | week 0, 12, 16
  The Quality of Life-Alzheimer's Disease (QOL-AD) has 13-items covering physical health, energy, mood, living situations, memory, family, marriage, friends, chores, fun, money, self and life as a whole. The QOL-AD uses straightforward language for simplicity, which will be conducted at baseline, 12 weeks, and follow-up (16 weeks).
Changes of Constitution in Chinese Medicine Questionnaire | week 0, 12, 16
  The Constitution in Chinese Medicine Questionnaire (CCMQ) consists of 60 items to classify a person into one or more of nine Body constitution(BC) types: gentleness (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). Coexistence of multiple imbalanced BC types was possible which is consistent with the TCM theories. The scoring algorithm proposed in the original CCMQ was adopted in this study. A higher score in the CCMQ BC scale indicates a higher likelihood of the specific BC type, and a score of 30 is set as threshold for case definition. The CCMQ will be conducted at baseline, 12 weeks, and follow-up (16 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan